CLINICAL TRIAL: NCT06179498
Title: A Randomized Trial to Test the Efficacy of a Partner Navigation Intervention for HCV Treatment Among Young Adult People Who Inject Drugs
Brief Title: Partner Navigation Intervention for Hepatitis C Treatment Among Young People Who Inject Drugs
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 1R01DA053325-01A1 (NIH); 1R01DA053325-01A1 (NIH)
Record Dates: First submitted 2023-12-12; First posted 2023-12-22 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Hepatitis C
Keywords: Young people who inject drugs
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Intervention Model Description: Behavioral intervention: two counseling based sessions
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): In addition to standard HCV results disclosure for the comparator arm, intervention participants will have two counseling sessions:
  Session 1: Immediately after HCV results disclosure, a staff-facilitated session with the index to (1) Establish HCV Treatment Goals, fostering commitment, and (2) Engage the Injecting Partner, identifying ways to support treatment initiation.
  Session 2: One week later, involving both the index and injecting partner, to (1) Enhance Partner Support with specific strategies for HCV treatment initiation and (2) Collaborative Navigation Mapping, using a "navigation map" tool. By Session 2's end, both will have a completed navigation map, a visual guide for the HCV treatment journey.
  Both sessions stress communication and dyadic coordination. The "navigation map" tool ensures a personalized plan for the index's treatment initiation and the partner's supportive navigator role.
  Interventions: Behavioral: Partner Navigation Intervention
- Control (No Intervention): Standard of care HCV disclosure. This staff-facilitated session follows the California HIV/HCV test counselor certification protocol with the Index alone.

INTERVENTIONS:
Behavioral: Partner Navigation Intervention — A two-session, disclosure counselor-led, behavioral intervention to enable the injecting partner to support and navigate the adult PWID to start HCV treatment.
  Arms: Intervention

SUMMARY:
The Partner Navigation Intervention Study is a randomized controlled study (RCT) to assess the efficacy and mechanism of action of the first behavioral intervention to increase hepatitis C (HCV) treatment initiation among adult people who inject drugs (PWID).

DETAILED DESCRIPTION:
After an initial ramp-up phase to ensure intervention materials and protocols meet the needs of the target population and organizational setting, we will apply a stratified randomized design to enroll 250 adult PWID with recently diagnosed HCV infection ("index") and their primary injecting partner("partner") into a randomized control efficacy trial of a two-session partner navigation intervention, compared to standard of care. The primary endpoint is starting HCV treatment. Recruitment will over sample PWID between 18-30 years of age.

ELIGIBILITY:
Inclusion Criteria:

* Self report injecting drugs in the past month
* Self report a primary injecting partner (currently inject drugs together)
* HCV infection identified at partnering community-based clinical site

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2024-03-25 (Actual); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Intervention efficacy | 6 months, 12 months, and 24 months after HCV infection disclosure visit.
  Assessed by comparing the proportion of those enrolled in the intervention group who initiated treatment to the proportion of those enrolled in the control group who initiated treatment at 6 months, 12 months, and 24 months after HCV infection disclosure visit.

SECONDARY OUTCOMES:
Change in Partner Support (Intervention mechanism) | 1 week, 1 month, 3 months and 6-months after HCV infection disclosure visit
  Self-reported level of partner support measured at baseline, 1 week, 1 month, 3 months, and 6 months. Partner support is measured with a validated survey scale (range 1-5) where the higher the value the higher the partner support.
HCV Treatment Completion | Point of HCV treatment initiation up to 3 years
  The proportion of participants who complete treatment, by randomized group
Sustained Virologic Response at 12 weeks post treatment completion (SVR12) | Point of HCV treatment initiation up to 3 years
  Proportion of participants who achieve sustained virologic response at 12 weeks post treatment (SVR12), by randomized group

CONTACTS AND LOCATIONS:
Overall Officials: Meghan D Morris, MPH, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Morris MD, Tan JY, McDonell CC, Scarpetta M, Nguyen TN, Price JC, Neilands TB. A single-site randomized controlled trial of partner navigation to HCV treatment for people who inject drugs: a study protocol for the You're Empowered for Treatment Initiation (YETI) partner trial. Trials. 2025 Jan 22;26(1):26. doi: 10.1186/s13063-024-08662-0. PMID 39844334